CLINICAL TRIAL: NCT01915576
Title: A Phase I, Multi-center, Non-randomized, Open-label, Dose Escalation Design Study to Characterize Safety, Tolerability, Pharmacokinetics and Maximum Tolerated Dose of BAY 1125976 in Subjects With Advanced Solid Tumors
Brief Title: Phase I Dose Escalation Study With an Allosteric AKT 1/2 Inhibitor in Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16447; 2012-004671-39 (EudraCT Number)
Record Dates: First submitted 2013-07-29; First posted 2013-08-05 (Estimated); Last update posted 2016-12-28 (Estimated); Status verified 2016-12

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- BAY1125976 [once daily, dose-esc.] (Experimental): Oral administration once daily. Starting dose is 10 mg and will be escalated depending on any dose-limiting toxicities
  Interventions: Drug: BAY1125976
- BAY1125976 [twice daily, dose-esc.] (Experimental): Oral administration twice daily. Starting dose is 40mg twice daily and will be escalated depending on any dose-limiting toxicities
  Interventions: Drug: BAY1125976
- BAY1125976 [MTD] (Experimental): Oral administration of the defined MTD which shows optimal safety, PK profile, PD target inhibition and preliminary efficacy (once daily or twice daily) in different patient groups
  Interventions: Drug: BAY1125976

INTERVENTIONS:
Drug: BAY1125976 — Oral administration once daily. Starting dose is 10 mg and will be escalated depending on any dose-limiting toxicities
  Arms: BAY1125976 [once daily, dose-esc.]
Drug: BAY1125976 — Oral administration twice daily. Starting dose is 40mg twice daily and will be escalated depending on any dose-limiting toxicities
  Arms: BAY1125976 [twice daily, dose-esc.]
Drug: BAY1125976 — Oral administration of the defined MTD which shows optimal safety, PK profile, PD target inhibition and preliminary efficacy (once daily or twice daily) in different patient groups
  Arms: BAY1125976 [MTD]

SUMMARY:
This is the first study where BAY1125976 is given to humans. Patients (all comers) will receive the study drug treatment in a dose-escalation scheme (no placebo group) to determine the safety, tolerability and maximum tolerated dose (MTD) of BAY1125976. The relative bioavailability of liquid service formulation and tablets will be determined.

After the MTD is defined breast cancer patients with and without AKT1 mutation will be treated.

The study will also assess the pharmacokinetics, biomarker status, pharmacodynamic parameters and tumor response of BAY1125976.

BAY1125976 will be given daily as single oral application. Treatment will be stopped if the tumor continues to grow, if side effects, which the patient cannot tolerate, occur or if the patient decides to exit treatment.

ELIGIBILITY:
Inclusion Criteria:

* For dose escalation cohorts: Subjects with advanced, histologically or cytologically confirmed solid tumors are eligible. Subjects' tumors (all comers) must be refractory to standard treatment with no standard therapy available, or subjects actively refuse any treatment, which would be regarded standard. In addition, the investigator must judge the experimental treatment as clinically and ethically acceptable
* For expansion cohort only: Subjects with histologically or cytologically proven metastatic breast cancer (with and without AKT1 E17K (G49A) mutation) or subjects with known AKT1 E17K (G49A) mutation in any other advanced solid tumor with at least one line of chemotherapy in the metastatic setting and not amenable to surgery with curative intent
* Subjects must have measurable disease (Response evaluation criteria in solid tumors (RECIST 1.1)
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0 - 2
* Bone marrow, liver and renal functions as assessed by adequate laboratory methods to be conducted within 7 days prior to starting study treatment
* Subjects must provide tumor biopsies before treatment
* Recovery to CTCAE (Common Terminology Criteria for Adverse Events Version 4.03) Grade 0 or Grade 1 or recovery to baseline preceding the prior treatment of any previous drug / procedure-related toxicity (except alopecia, anemia, and hypothyroidism)

Exclusion Criteria:

* History of cardiac disease including congestive heart failure > New York Heart Association (NYHA) Class II
* Subjects with type 1 or type 2 diabetes mellitus
* Subjects with fasting glucose >125 mg/dL in 2 independent measurements or glycated hemoglobin (HbA1c) ≥ 7%
* Moderate and severe hepatic impairment, i.e. Child-Pugh B or C
* Active infections of CTCAE (Common Terminology Criteria for Adverse Events Version 4.03) Grade >2 or infections of CTCAE Grade 2 not responding to therapy
* Symptomatic metastatic brain or meningeal tumors unless the patient is > 3 months from definitive therapy, has a negative imaging study within 4 weeks of study entry and is clinically stable with respect to the tumor at the time of study entry.
* Subjects undergoing renal dialysis
* Previous or concurrent cancer that is distinct in primary site or histology from the cancer being evaluated in this study except cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors (Ta, Tis & T1) or any cancer curatively treated > 3 years prior to study entry
* Autologous bone marrow transplant or stem cell rescue within 4 months of study entry
* Treatment with oral steroids (dose ≥ 10 mg/day of methylprednisolone or equivalent)
* Clinically relevant findings in the ECG such as a second- or third-degree AV block, prolongation of the QRS complex over 120 msec or of the QTcF-interval over 450 msec
* Acute toxic effects of previous anticancer chemotherapy or immunotherapy have to be normalized to CTCAE Grade equal or lower than 1 (excluding alopecia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2013-09; Primary Completion 2016-07 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability | up to 2 years
Maximum tolerated dose (MTD) of BAY1125976 | up to 2 years
Area under the plasma concentration vs time curve from zero to infinity after single (first) dose | at pre-dose and 0.5, 1, 2, 4, 6, 8, 12 and 24 hours post-dose

SECONDARY OUTCOMES:
Food effect assessment | up to 2 years
  The effect of a high-fat, high-calorie meal on the pharmacokinetic parameters of BAY1125976 will be determined in 6 - 9 subjects in the MTD dose level or a lower dose level receiving the tablet for the cohort of the dose escalation part.
Tumor response will be evaluated based on Response Evaluation Criteria in Solid Tumors (RECIST) definitions | up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (7):
- United States (4):
  - Santa Monica, California
  - Boston, Massachusetts
  - St Louis, Missouri
  - Houston, Texas
- Villejuif, France
- Heidelberg, Baden-Wurttemberg, Germany
- Sankt Gallen, Canton of St. Gallen, Switzerland